CLINICAL TRIAL: NCT00339404
Title: Genetic Analysis of Familial Melanoma
Status: Completed | Type: Observational
Sponsor: National Human Genome Research Institute (NHGRI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999999012; OH99-HG-N012
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2011-03-07

CONDITIONS: Melanoma
Keywords: Genotyping; Linkage Analysis; Cancer; Hereditary Melanoma
MeSH Terms: conditions — Melanoma; Neoplasms; Melanoma, Cutaneous Malignant

SUMMARY:
In collaboration with members of The International Melanoma Consortium, we propose to study melanoma in families lacking mutations in the cyclin-dependent kinase inhibitor 2 (CDKN2 or p16) gene, or the cyclin-dependant kinase 4 (CDK4). CDKN2 and CDK4 are both genes that encode presumed tumor suppressor genes, mutant forms of which are known to cause increased susceptibility to melanoma. The purpose of the present study then is to confirm the existence of and to identify additional gene(s) involved in heritable melanoma (cutaneous and ocular) and their precursor lesions (atypical nevi) by linkage analysis and gene mapping strategies. It is clear that the risk to develop atypical nevi and/or melanoma is strongly influenced by genetic and environmental factors (e.g. sun exposure). Characterization of such genes could provide important insights into the inheritance, pathogenesis, and treatment of this increasingly important disease.

DETAILED DESCRIPTION:
In collaboration with members of The International Melanoma Genetics Consortium, we propose to study melanoma in families lacking mutations in the cyclin-dependent kinase inhibitor 2 (CDKN2A), or the cyclin-dependant kinase 4 (CDK4) genes. CDKN2 and CDK4 are both genes that encode presumed tumor suppressor genes, mutant forms of which are known to cause increased susceptibility to melanoma. The purpose of the present study then is to confirm the existence of and to identify additional gene(s) involved in heritable melanoma (cutaneous and ocular) and their precursor lesions (atypical nevi) by linkage analysis and gene mapping strategies. It is clear that the risk to develop atypical nevi and/or melanoma is strongly influenced by genetic and environmental factors (e.g. sun exposure). Characterization of such genes could provide important insights into the inheritance, pathogenesis, and treatment of this increasingly important disease.

ELIGIBILITY:
* INCLUSION CRITERIA:

Inclusion into this study was restricted to families containing at least three CMM cases with DNA available for genotyping, and CDKN2A and CDK4 involvement and had been excluded.

All families must be mutation negative for both CDKN2A and CDK4.

This study will also include families with at least one case of ocular and two cases of other cutaneous melanomas, or at least 2 ocular melanomas (except where they occur in parent and child).

EXCLUSION CRITERIA:

Any family showing evidence of haplotype sharing in the 9p21-p22 region, where CDKN2A is located, was also excluded.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3000 (Estimated)
Dates: Start 1999-03-04; Study Completion 2011-03-07

CONTACTS AND LOCATIONS:
Locations (1):
- National Human Genome Research Institute (NHGRI), 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Hussussian CJ, Struewing JP, Goldstein AM, Higgins PA, Ally DS, Sheahan MD, Clark WH Jr, Tucker MA, Dracopoli NC. Germline p16 mutations in familial melanoma. Nat Genet. 1994 Sep;8(1):15-21. doi: 10.1038/ng0994-15. PMID 7987387
- [Background] Kamb A, Shattuck-Eidens D, Eeles R, Liu Q, Gruis NA, Ding W, Hussey C, Tran T, Miki Y, Weaver-Feldhaus J, et al. Analysis of the p16 gene (CDKN2) as a candidate for the chromosome 9p melanoma susceptibility locus. Nat Genet. 1994 Sep;8(1):23-6. doi: 10.1038/ng0994-22. PMID 7987388
- [Background] Hayward NK. The current situation with regard to human melanoma and genetic inferences. Curr Opin Oncol. 1996 Mar;8(2):136-42. doi: 10.1097/00001622-199603000-00011. PMID 8727306